CLINICAL TRIAL: NCT00355199
Title: Multicentric Randomized Phase III Study Comparing High Doses of Chemotherapy With Rituximab Followed by Auto-transplant HPC Versus CHOP Plus Rituximab as First Line Therapy in High Risk Patients With DLBCL Non-Hodgkin's Lymphomas
Brief Title: Comparison of HD Chemotherapy Followed by Auto-transplant and R-CHOP in High Risk Patients With DLBCL.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Terapie Innovative nei Linfomi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT: 2005-00700-14
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; R-HDS; R-CHOP14
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-HDS (Experimental): R-HDS : Rituximab supplemented high-dose (Cyclophosphamide,Ara-C, Methotrexate, Etoposide, Cis-Platin) sequential chemotherapy with autografting.
  Interventions: Drug: Rituximab-HDS
- R-CHOP (Active Comparator): Rituximab-CHOP (cyclophosphamide/doxorubicin/vincristine/prednisone).
  Interventions: Drug: Rituximab-CHOP

INTERVENTIONS:
Drug: Rituximab-HDS — Rituximab-HDS
  Other Names: Rituximab supplemented high-dose sequential chemotherapy.
  Arms: R-HDS
Drug: Rituximab-CHOP — Rituximab-CHOP
  Other Names: Rituximab/Cyclophosph/doxorubic/vincrist/prednis
  Arms: R-CHOP

SUMMARY:
Multicentric randomized phase III study comparing high doses of chemotherapy with Rituximab followed by auto-transplant HPC versus CHOP plus Rituximab as first line therapy in high risk patients with DLBCL Non-Hodgkin's lymphomas.

DETAILED DESCRIPTION:
Diffuse large B cells Non-Hodgkin's lymphomas represents one of the most frequent form of lymphoma. Its clinical development progresses rapidly and is characterized by a biphasic survival curve with patients in complete remission (which can be considered cured) and patients that relapse. This last group of subjects have only 25%-33% chance of long free disease survival if treated with a second line therapy with high dose chemotherapy plus autologous transplant of PBPC.

Therefore in order to achieve an improvement of the overall survival in patient with DLBCL, it is necessary to increase the number of complete remission after first line therapy.

The aim of R-HDS study, multicentre randomized phase III trial, is to evaluate and compare the efficacy and safety of an intensive conditioning regimen with high intensity chemo-immunotherapy (R-HDS) plus autologous transplantation versus CHOP conditioning regimen plus Rituximab in patients with unfavorable prognosis at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DLBCL CD20+.
* Patients with Ann Arbor classification B-bulk >= II
* Patients of age between 18-65 with age-adjusted IPI 2-3 and ECOG performance status 0-3 or patients of age 61-65 with IPI 3, 4, 5 and ECOG performance status 0-2. The disease stage criteria must be documented with instrumental examinations and bone marrow biopsy.
* Hematology parameters one week before starting study as follows: Hb >= 9 g/dl, WBC >= 3 x 10exp9/l, neutrophils >= 1.5 x 10exp9/l, PLT >= 100 x 10exp9/l.
* Patients with pulmonary DLCO >= 50% and cardiac EF >= 40%.
* Voluntary written informed consent must be signed before recruitment, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care. Patients must to be informed on the risk of sterility and they must agree to use contraception for the duration of the study. Male subject have to the opportunity of freezing seminal fluid.

Exclusion Criteria:

* Diagnosis different from that describe above.
* Patients with concomitant, serious and uncontrolled illnesses such as cardiopathies (i.e. congestive cardiopathy, ischemic hearth disease, cardiac arrhythmia not controlled by therapy, IMA in the last six months, hearth disease NYHA class III or IV), hepatopathy not related to the lymphoma (bilirubin >= 2 mg/dl, ALT >= 2.5 times the normal value, alkaline phosphatase >=2.5 times the upper limit), kidneys insufficiency not related to the lymphoma (creatinine >=2 mg/dl).
* Patients affected by opportunistic infections or with positive serology for HIV, HCV, HbsAg (cases with normal levels of hepatic enzymes and not showing active viral replication documented with HBV-DNA are not excluded from randomization; patients with HBV+ can be enrolled after receiving prophylaxis with lamivudina one week before starting chemotherapy. These patients should be monitored twice a month for HbsAg, HBCab, HBV-DNA).
* Patients which have or have had another type of cancer exception made for skin cancers (melanoma and "in situ" cervical cancer not included).
* Patient with a history of anaphylaxes or more generally patients which have had any serious allergic reaction after serum infusion.
* Patient with uncontrolled epilepsy, CNS disorders or psychiatric problems which, according to the investigator, is likely to interfere with participation in this clinical study (i.e. the signing of the informed consent, therapy compliance).
* Inability to attend follow-up visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2005-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cortelazzo, MD, Study Chair — Divisione di Ematologia - Ospedale Centrale di Bolzano - 39100 Bolzano Italy
Locations (16):
- Italy (16):
  - Clinica di Ematologia - Nuovo Ospedale Torrette, Ancona
  - U.O. Ematologia - Ospedali Riuniti di Bergamo, Bergamo
  - Divisione di Ematologia - Ospedale Centrale di Bolzano, Bolzano
  - CTMO - Ematologia - Ospedale "R. Binaghi", Cagliari
  - Divisione di Ematologia - Ospedale Ferrarotto, Catania
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Divisione Ematologia - Istituto S. Raffaele, Milan
  - Oncologia Medica - Istituto Nazionale dei Tumori, Milan
  - U.O. Ematologia - Istituto Nazionale dei Tumori, Milan
  - Divisione di Ematologia - Azienda Ospedaliera, Padua
  - Ematologia - Azienda Ospedaliera V. Cervello, Palermo
  - Ematologia Clinica - Ospedale Civile di Pescara, Pescara
  - Ematologia e TMO - Ospedale S. Camillo, Roma
  - Divisione Universitaria di Ematologia - Azienda Ospedaliera S. Giovanni Battista (Molinette), Torino
  - Dipartimento di Medicina Clinica e Sperimentale - Università di Verona, Verona
  - Divisione di Ematologia - Presidio Ospedaliero S. Bortolo, Vicenza

REFERENCES:
- [Derived] Derenzini E, Mazzara S, Melle F, Motta G, Fabbri M, Bruna R, Agostinelli C, Cesano A, Corsini CA, Chen N, Righi S, Sabattini E, Chiappella A, Calleri A, Fiori S, Tabanelli V, Cabras A, Pruneri G, Vitolo U, Gianni AM, Rambaldi A, Corradini P, Zinzani PL, Tarella C, Pileri S. A three-gene signature based on MYC, BCL-2 and NFKBIA improves risk stratification in diffuse large B-cell lymphoma. Haematologica. 2021 Sep 1;106(9):2405-2416. doi: 10.3324/haematol.2019.236455. PMID 32817282

RESULTS

PARTICIPANT FLOW:
Groups:
- R-HDS: R-HDS: 3 APO: first Doxorubicin at 50 mg/m2 iv, then at 75 mg/m2 iv days 14, 28; Vincristine 1.4 mg/m2 iv days 1,14,28; Prednisone p.o 40 mg/m2 days1-28). Subsequently:high-dose (hd) Cyclophosphamide 7 g/m2 iv, day 1+ Rituximab 375 mg/m2 iv days +3;+11, harvest of peripheral blood progenitor cells (PBPC); hd-Cytarabine 2 g/m2 iv bid for 6 days. Day 7:infusion 1.5-2x10^6 autologous CD34+ cells/kg, Rituximab 375 mg/m2 iv day+8;+16; hd-Etoposide 2.4 g/m2 iv day +1, Cisplatin 100 mg/m2 iv day+2; PBPC (2x10^6 CD34+ cells/Kg) reinfused following etoposide/cisplatin. ASCT conditioned with mitoxantrone 60 mg/m2 iv day -5 and melphalan 180 mg/m2 iv day -2 or BEAM (BCNU 300 mg/m2 iv day -6, Etoposide 200 mg/m2 iv days -5 to -2, Ara-C 200 mg/m2 iv every 12 h x8 doses, days from -5 to -2, Melphalan 140 mg/m2 iv day-1),supported by PBPC autograft day 0. Two Rituximab days +14;+24 after ASCT. Patients with initial bulky or residual lesions received IFRT within 2-3 months after chemotherapy program.
- R-CHOP 14: Patients enrolled into the control arm R-CHOP (rituximab 375 mg/m2 i.v., cyclophosphamide 750 mg/m2 i.v., doxorubicin 50 mg/m2 i.v., vincristine 1.4 mg/m2 i.v. given on day 1 and 100 mg/d of prednisone p.o. on days 1-5), given every 14 days x 8 cycles. The neutropenic phase was supported by G-CSF (filgrastrim 5μg/kg s.c. daily or Pegfilgrastim s.c. given once on day +1 of each cycle). CNS prophylaxis with intrathecal chemotherapy (MTX, ARAC, steroids) was given to high risk patients who, at diagnosis, had infiltration of the bone marrow, testes, Waldeyer ring, cranial air sinuses (including nasal), salivary glands and epidural space. In R-CHOP, 33 patients (27%) received intrathecal prophylaxis. Patients with initial bulky or residual lesions received IFRT within 2-3 months after chemotherapy program.
Period: Overall Study
Arm/Group | R-HDS | R-CHOP 14
Started | 120 | 126
Completed | 113 | 122
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R-HDS | R-CHOP | Total
Number analyzed (Participants) | 113 | 122 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 113 | 120 | 233
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 51 | 99
  Male | 65 | 71 | 136
Region of Enrollment [Number; unit: participants]
  Italy | 113 | 122 | 235

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival
Description: EFS was defined from the time of the study entry to any treatment failure including disease progression or discontinuation of treatment for any reason or date of the last follow-up visit
Time Frame: 36 months from end of therapy
Measure: Number (95% Confidence Interval); unit: percentage of EFS at 3 years follow-up
Groups:
- R-HDS: Patients treated with high dose sequential chemotherapy program (R-HDS) with ASCT.
- R-CHOP 14: Patients treated with R-CHOP-14 (8 cycles)
Arm/Group | R-HDS | R-CHOP 14
Number analyzed (Participants) | 113 | 122
percentage of EFS at 3 years follow-up | 65 [56 to 74] | 62 [54 to 71]
Statistical Analysis 1: Comparison: R-HDS vs R-CHOP 14; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.66 to 1.48] — HR refers to R-HDS (R-CHOP is the reference level)

2. Secondary Outcome: Complete Remission
Description: Clinical response was assessed by complete restaging according to Cheson criteria. Cheson BD, Pfistner B, Juweid ME, et al: Revised response criteria for malignant lymphoma. J Clin Oncol 25:579-86, 2007
Time Frame: Through therapy completion an average of 8 months
Measure: Number; unit: participants
Arm/Group | R-HDS | R-CHOP 14
Number analyzed (Participants) | 113 | 122
participants | 86 | 95

3. Secondary Outcome: Disease Free Survival
Description: DFS was defined from the time of documentation of CR to time to relapse or death as a result of lymphoma or acute toxicity of treatment or date of the last follow-up visit
Time Frame: 36 months from end of therapy
Measure: Number (95% Confidence Interval); unit: percentage of DFS at 3 years follow-up
Arm/Group | R-HDS | R-CHOP 14
Number analyzed (Participants) | 86 | 95
percentage of DFS at 3 years follow-up | 91 [85 to 97] | 79 [71 to 87]
Statistical Analysis 1: Comparison: R-HDS vs R-CHOP 14; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.29 to 1.21] — HR refers to R-HDS (R-CHOP is the reference level)

4. Secondary Outcome: Overall Survival
Description: OS was defined from the time of the study entry to death as a result of any cause or date of the last follow-up visit
Time Frame: 36 months from end of therapy
Measure: Number (95% Confidence Interval); unit: percentage of OS at 3 years follow-up
Arm/Group | R-HDS | R-CHOP 14
Number analyzed (Participants) | 113 | 122
percentage of OS at 3 years follow-up | 77 [70 to 86] | 74 [67 to 82]
Statistical Analysis 1: Comparison: R-HDS vs R-CHOP 14; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.57 to 1.52] — HR refers to R-HDS (R-CHOP is the reference level)

5. Secondary Outcome: Toxicity
Description: Percentage of participants with at least one reported episode of CTC grade III or IV toxic events
Time Frame: Through therapy completion an average of 8 months
Measure: Number; unit: percentage of participants
Arm/Group | R-HDS | R-CHOP 14
Number analyzed (Participants) | 113 | 122
percentage of participants
  Grade III or IV Neutropenia | 84 | 34
  Grade III or IV Anemia | 71 | 15
  Grade III or IV Thrombocytopenia | 86 | 5
  Grade III or IV Gastrointestinal | 29 | 11
  Grade III or IV Cardiac | 4 | 7
  Grade III or IV Neurological | 0 | 7
  Grade III or IV Hepatic and Metabolic | 7 | 6
  Grade III or IV Infection | 54 | 8

6. Secondary Outcome: Efficacy of R-HDS Conditioning as Salvage Therapy in Patients Non-responders After Four Cycles of R-CHOP 14
Time Frame: Through completion of salvage therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through therapy scheduled and follow-up completion
Description: Adverse event is any undesirable medical event (symptom or illness, including any abnormal laboratory values), which occurred during treatment or during the follow-up period, regardless of its relationship to treatment in use.
  Were reported Adverse events with severity > 2
Arm/Group | R-HDS | R-CHOP 14
All-Cause Mortality (participants affected / at risk) | 30/113 | 35/122
Serious Adverse Events (participants affected / at risk) | 29/113 | 10/122
Other Adverse Events (participants affected / at risk) | 0/113 | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-HDS (N=113) | R-CHOP 14 (N=122)
Infection (Infections and infestations) | 16 (28) | 4 (6)
Blood/bone marrow cellularity (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cardiac (Cardiac disorders) | 3 (3) | 0 (0)
Neurology (Nervous system disorders) | 2 (2) | 1 (1)
Hemorrhage/bleeding (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Renal (Renal and urinary disorders) | 2 (2) | 0 (0)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vascular (Vascular disorders) | 1 (1) | 0 (0)
Death (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No